CLINICAL TRIAL: NCT01431079
Title: Designing and Evaluating a Health Belief Model Based Intervention to Increase Intent of HPV Vaccination Among College Men: Use of Qualitative and Quantitative Methodologies
Brief Title: A Health Belief Model Based Intervention to Increase Human Papilloma Virus (HPV) Vaccination Among College Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Sharma Manoj, Professor, University of Cincinnati
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 11083108; 39991 (Other: Merck Pharmaceuticals)
Record Dates: First submitted 2011-09-03; First posted 2011-09-09 (Estimated); Results first posted 2012-12-10 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: HPV Vaccine Acceptability
Keywords: HPV; College men; HPV vaccine; Health belief model; HPV vaccine acceptance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health belief model based education (Experimental): This experimental arm will provide an educational intervention designed to modify constructs of health belief model regarding HPV vaccine acceptability.
  Interventions: Behavioral: HPV vaccine acceptability
- Knowledge-based education (Active Comparator): This comparison arm will provide education based on knowledge regarding HPV vaccine acceptability.
  Interventions: Behavioral: HPV vaccine acceptability

INTERVENTIONS:
Behavioral: HPV vaccine acceptability — One arm will receive health belief model based educational intervention and other arm will receive knowledge-based educational intervention.

SUMMARY:
The purposes of this study are to (1) identify predictors of Human papillomavirus (HPV) vaccine acceptability among college men based on the Health Belief Model through focus groups, (2) triangulate focus group results with a prior quantitative study in developing an intervention based on the Health Belief Model to enhance HPV vaccine acceptability, and (3) test the efficacy of the above intervention based on the Health Belief Model by comparing it to a knowledge-based intervention. Approximately five focus groups with ten participants in each group with college students in the ages 18-25 years will be conducted at a large Midwestern University for the qualitative piece. Data will be analyzed for categories and triangulated with previous study to develop a theory based intervention. For the quantitative piece a randomized controlled design with 45 participants in each arm (theory based intervention and knowledge based intervention) will be implemented.

DETAILED DESCRIPTION:
Up to this date, there was a lack of qualitative research on vaccine acceptability among men and theory-based interventions that promote HPV vaccination among men. A few studies have been conducted with parents and physicians regarding HPV vaccination with girls, and a few regarding women's awareness and acceptability. Results indicated increasing awareness of HPV, informing costs and benefits associated with the vaccine, and perceived susceptibility. Based on this information, it is crucial to obtain a further understanding of knowledge, awareness, and predictors related to HPV and its vaccination in men. Information obtained can be utilized in developing an intervention to increase intentions of taking the HPV vaccine. Refining results will lead to a standardization of an intervention that can be implemented across college campuses.

ELIGIBILITY:
Inclusion Criteria:

* Males
* English speaking
* 18-25 years
* Undergraduate or graduate student at the University of Cincinnati

Exclusion Criteria:

* Females
* Under 18 years, or above 25 years
* Non- English speaking individuals
* Non-university attending students
* If already received HPV vaccination

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Sharma, Ph.D., Principal Investigator — University of Cincinnati; Rebecca Lee, Ph.D., Study Director — University of Cincinnati; Purvi Mehta, MS, Study Director — University of Cincinnati
Locations (1):
- Manoj Sharma, Cincinnati, Ohio, United States

REFERENCES:
- See also: Manufactures HPV vaccine — http://www.merck.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for Phase I of the study was conducted between Oct. 2011-Nov. 2011 at the University of Cincinnati. Snowball sampling was done (n=50).
  Phase II occurred between March 2012-April 2012 at the University. A snowball sample was used. 90 participants were recruited. A post test was done immediately after the intervention.
Groups:
- Health Belief Model Based Education: This experimental arm will provide an educational intervention designed to modify constructs of health belief model regarding HPV vaccine acceptability.
  HPV vaccine acceptability : One arm will receive health belief model based educational intervention and other arm will receive knowledge-based educational intervention.
- Knowledge-based Education: This comparison arm will provide education based on knowledge regarding HPV vaccine acceptability.
  HPV vaccine acceptability : One arm will receive health belief model based educational intervention and other arm will receive knowledge-based educational intervention.
Period: Overall Study
Arm/Group | Health Belief Model Based Education | Knowledge-based Education
Started | 45 | 45
Post-test | 45 | 45
Completed | 10 | 6
Not Completed | 35 | 39
Not completed — Lost to Follow-up | 35 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Belief Model Based Education | Knowledge-based Education | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 45 | 90
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 19.76 (1.04) | 20.6 (2.44) | 20.2 (1.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 45 | 45 | 90
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Post Intervention to Follow-up (up to 3 Months) After the Interventions the Number of Participants Who Have Taken the HPV Vaccine
Description: Before, after and one to three month following the health belief model based educational intervention and knowledge-based educational intervention the participants will be asked if they have taken the first dose of HPV vaccine and changes noted.
Time Frame: Post intervention and up to 3 months after the interventions
Population: A sample size of 90 men total (Erdfleder, Faul, & Buchner, 1996) was needed for the intervention. This was calculated by G*Power based on: alpha= 0.05, power=.80, groups=2, measurements=2, effect size=.20, correlations among repeated measures-0.5, nonsphericity correction ε=1, giving us total sample of 90.
Measure: Number; unit: participants
Groups:
- Baseline Health Belief Model Based Education: This experimental arm will provide baseline data for number of people who have taken HPV vaccine before an educational intervention designed to modify constructs of health belief model regarding HPV vaccine acceptability.
  HPV vaccine acceptability : One arm will receive health belief model based educational intervention and other arm will receive knowledge-based educational intervention.
- Baseline Knowledge-based Education: This comparison arm will provide baseline data for number of people who have taken the HPV vaccine before an education based on knowledge regarding HPV vaccine acceptability.
  HPV vaccine acceptability : One arm will receive health belief model based educational intervention and other arm will receive knowledge-based educational intervention.
- Post Test Health Belief Model Based Education: This experimental arm will provide post test data for number of people who have taken HPV vaccine after an educational intervention designed to modify constructs of health belief model regarding HPV vaccine acceptability.
- Post Test Knowledge-based Education: This comparison arm will provide post test data for number of people who have taken the HPV vaccine after an education based on knowledge regarding HPV vaccine acceptability.
- Follow-up Health Belief Model Based Education: This experimental arm will provide follow-up data for number of people who have taken HPV vaccine upto 3 months after an educational intervention designed to modify constructs of health belief model regarding HPV vaccine acceptability.
- Follow-up Knowledge-based Education: This comparison arm will provide follow-up data for number of people who have taken the HPV vaccine after an education based on knowledge regarding HPV vaccine acceptability.
Arm/Group | Baseline Health Belief Model Based Education | Baseline Knowledge-based Education | Post Test Health Belief Model Based Education | Post Test Knowledge-based Education | Follow-up Health Belief Model Based Education | Follow-up Knowledge-based Education
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 10 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline to Post Intervention to Follow-up up to 3 Months After the Interventions the Number of Participants Who Intend to Take HPV Vaccine Using HPV Intent Scale (Possible Range 0-4 Likert Units)
Description: Before the interventions, post test after the interventions and follow-up 1 to 3 months after the interventions (health belief model based and knowledge based) participants will be asked about their intent to take the HPV vaccine on a scale of 0-4 Likert units and changes noted.
  Posttest was conducted immediately after the intervention. Minimum score = 0 indicating no intent to take vaccine; Maximum score = 4 indicating strong intent to take vaccine. Scale was a single item scale.
Time Frame: Post intervention and up to 3 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline Health Belief Model Based Education: This experimental arm will provide baseline data for an educational intervention designed to modify constructs of health belief model regarding HPV vaccine acceptability.
  HPV vaccine acceptability : One arm will receive health belief model based educational intervention and other arm will receive knowledge-based educational intervention.
- Baseline Knowledge-based Education: This comparison arm will provide baseline data regarding education based on knowledge regarding HPV vaccine acceptability.
  HPV vaccine acceptability : One arm will receive health belief model based educational intervention and other arm will receive knowledge-based educational intervention.
- Post Test Health Belief Model Based Education: This experimental arm will provide post test data for an educational intervention designed to modify constructs of health belief model regarding HPV vaccine acceptability.
- Post Test Knowledge Based Education: This comparison arm will provide post test data regarding education based on knowledge regarding HPV vaccine acceptability.
- Follow-up Health Belief Model Based Education: This experimental arm will provide follow-up data for an educational intervention designed to modify constructs of health belief model regarding HPV vaccine acceptability.
- Follow-up Knowledge Based Education: This comparison arm will provide follow-up data regarding education based on knowledge regarding HPV vaccine acceptability.
Arm/Group | Baseline Health Belief Model Based Education | Baseline Knowledge-based Education | Post Test Health Belief Model Based Education | Post Test Knowledge Based Education | Follow-up Health Belief Model Based Education | Follow-up Knowledge Based Education
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 10 | 6
units on a scale | 2.16 (1.13) | 2.28 (1.14) | 2.78 (1.11) | 2.27 (1.10) | 2.70 (1.06) | 1.67 (1.03)

3. Secondary Outcome: Change From Baseline to Post Intervention to Follow-up (up to 3 Months) After the Interventions in Score of Perceived Susceptibility for HPV
Description: Before the interventions, after the interventions and up to 3 months following the interventions the health belief model construct of perceived susceptibility for HPV scores will be measured on a paper pencil self-report test and changes noted. Perceived susceptibility for HPV will be measured as a summative score on a three item Likert subscale with a range of 0 to 12 (0- not likely and 12-very likely). The subscale has acceptable validity and reliability.
  Difference between posttest and pre-test was done. This value was then used to run the multiple regressions.
Time Frame: Post interventions and up to 3 months after the interventions
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline Knowledge-based Education: This comparison arm will provide baseline data for education based on knowledge regarding HPV vaccine acceptability.
  HPV vaccine acceptability : One arm will receive health belief model based educational intervention and other arm will receive knowledge-based educational intervention.
- Post Test Health Belief Model Based Education: This experimental group will provide post test data for an HBM based educational intervention designed to modify constructs of health belief model regarding HPV vaccine acceptability.
- Post Test Knowledge Based Education: This control group will provide post test data for knowledge based education for HPV vaccine
- Follow-up Health Belief Model Based Education: This experimental group will provide follow-up data for an Health belief model based educational intervention designed to modify constructs of health belief model regarding HPV vaccine acceptability.
- Follow-up Knowledge Based Education: This control group will provide follow-up data for knowledge based education for HPV vaccine
Arm/Group | Baseline Health Belief Model Based Education | Baseline Knowledge-based Education | Post Test Health Belief Model Based Education | Post Test Knowledge Based Education | Follow-up Health Belief Model Based Education | Follow-up Knowledge Based Education
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 10 | 6
units on a scale | 3.69 (2.82) | 3.51 (3.00) | 5.84 (3.65) | 3.67 (2.99) | 4.80 (3.62) | 5.67 (3.78)

4. Secondary Outcome: Change From Baseline to Post Test to Upto 3 Month Follow-up After the Interventions in Score for Perceived Severity for HPV
Description: Before the interventions, after the interventions and up to 3 months following the interventions the health belief model construct of perceived severity for HPV scores will be measured on a paper pencil self-report test and changes noted. Perceived severity for HPV will be measured as a summative score on a three item Likert subscale with a range of 0 to 12 to 12 (0- not likely and 12-very likely). The subscale has acceptable validity and reliability.
  Difference between posttest and pre-test was done. This value was then used to run the multiple regressions.
Time Frame: Post interventions and up to 3 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline Health Belief Model Based Education: This experimental arm will provide base line data for an educational intervention designed to modify constructs of health belief model regarding HPV vaccine acceptability.
  HPV vaccine acceptability : One arm will receive health belief model based educational intervention and other arm will receive knowledge-based educational intervention.
- Post Test Knowledge Based Education: This comparison arm will provide post test data for education based on knowledge regarding HPV vaccine acceptability.
- Follow-up Knowledge Based Education: This comparison arm will provide follow-up data for education based on knowledge regarding HPV vaccine acceptability.
Arm/Group | Baseline Health Belief Model Based Education | Baseline Knowledge-based Education | Post Test Health Belief Model Based Education | Post Test Knowledge Based Education | Follow-up Health Belief Model Based Education | Follow-up Knowledge Based Education
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 10 | 6
units on a scale | 9.22 (1.93) | 9.06 (1.85) | 10.44 (1.62) | 9.11 (1.79) | 11.10 (1.37) | 8.83 (3.37)

5. Secondary Outcome: Change From Baseline to Post Test After the Interventions to up to 3 Month Follow-up in Score of Perceived Benefits of HPV Vaccine
Description: Before the interventions, after the interventions and one month following the interventions the health belief model construct of Perceived benefits of HPV vaccine scores will be measured on a paper pencil self-report test and changes noted. Perceived benefits of HPV vaccine will be measured as a summative score on a four item Likert subscale with a range of 0 to 16 (0-not very likely and 16- very likely). The subscale has acceptable validity and reliability.
  Difference between posttest and pre-test was done. This value was then used to run the multiple regressions.
Time Frame: post intervention and up to 3 months after the interventions
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline Knowledge-based Education: This comparison arm will provide baseline data for an education based on knowledge regarding HPV vaccine acceptability.
  HPV vaccine acceptability : One arm will receive health belief model based educational intervention and other arm will receive knowledge-based educational intervention.
- Post Test Health Belief Model Based Education: This experimental arm will provide posttest data for an educational intervention designed to modify constructs of health belief model regarding HPV vaccine acceptability.
- Post Test Knowledge-based Education: This comparison arm will provide post test data for an education based on knowledge regarding HPV vaccine acceptability.
- Follow-up Knowledge Based Education: This comparison arm will provide follow-up data for an education based on knowledge regarding HPV vaccine acceptability.
Arm/Group | Baseline Health Belief Model Based Education | Baseline Knowledge-based Education | Post Test Health Belief Model Based Education | Post Test Knowledge-based Education | Follow-up Health Belief Model Based Education | Follow-up Knowledge Based Education
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 10 | 6
units on a scale | 5.76 (1.59) | 7.08 (2.05) | 9.04 (1.02) | 7.40 (2.13) | 7.90 (1.97) | 5.67 (1.86)

6. Secondary Outcome: Change From Baseline to Post Test After the Interventions to Follow-up (up to 3 Months) in the Score of Perceived Barriers to Receiving HPV Vaccine
Description: Before the interventions, post test after the interventions following the interventions the health belief model construct of perceived barriers to receiving HPV vaccine scores will be measured on a paper pencil self-report test and changes noted. Perceived barriers for receiving HPV vaccine will be measured as a summative score on a three item Likert subscale with a range of 0 to 12 (0- not likely to 12- very likely). The subscale has acceptable validity and reliability.
  A difference between post-test and pre-test were taken to obtain the score. This score was then used in the regression.
Time Frame: post interventions and up to 3 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Post Test Knowledge-based Education: This comparison arm will provide post test data for education based on knowledge regarding HPV vaccine acceptability.
- Follow-up Knowledge-based Education: This comparison arm will provide follow-up data for education based on knowledge regarding HPV vaccine acceptability.
Arm/Group | Baseline Health Belief Model Based Education | Baseline Knowledge-based Education | Post Test Health Belief Model Based Education | Post Test Knowledge-based Education | Follow-up Health Belief Model Based Education | Follow-up Knowledge-based Education
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 10 | 6
units on a scale | 6.58 (1.95) | 5.35 (1.92) | 3.53 (2.04) | 5.49 (1.89) | 4.30 (2.98) | 6.50 (1.98)

7. Secondary Outcome: Change From Baseline to After the Interventions to Follow-up up to 3 Months After the Interventions in Score of Cues to Action to Receiving HPV Vaccine
Description: Before the interventions, and after the interventions and up to 3 months after the interventions the health belief model construct of cues to action to receiving HPV vaccine scores will be measured on a paper pencil self-report test and changes noted. Cues to action to receiving HPV vaccine will be measured as a summative score on a four item Likert subscale with a range of 0 to 16 (0- not at all likely to 16-very likely). The subscale has acceptable validity and reliability.
  Difference between post and pre-test were used to obtain a change score. This score was used for regressions.
Time Frame: Post interventions and up to three months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline Health Belief Model Based Education | Baseline Knowledge-based Education | Post Test Health Belief Model Based Education | Post Test Knowledge-based Education | Follow-up Health Belief Model Based Education | Follow-up Knowledge Based Education
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 10 | 6
units on a scale | 3.44 (2.73) | 4.35 (2.72) | 5.07 (2.78) | 4.27 (2.57) | 6.50 (3.17) | 6.67 (5.09)

8. Secondary Outcome: Change From Baseline and After the Interventions to up to 3 Months Follow-up in Score of Self-efficacy for Receiving HPV Vaccine
Description: Before the interventions and after the interventions the health belief model construct of self-efficacy for receiving HPV vaccine scores will be measured on a paper pencil self-report test and changes noted. Self-efficacy for receiving HPV vaccine will be measured as a summative score on a three item Likert subscale with a range of 0 to 12 (0- not likely to 12- very likely). The subscale has acceptable validity and reliability.
  The difference between post and pre-test was taken to determine a change score. This score was then used for regressions.
Time Frame: Post interventions and up to 3 months follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline Health Belief Model Based Education | Baseline Knowledge-based Education | Post Test Health Belief Model Based Education | Post Test Knowledge-based Education | Follow-up Health Belief Model Based Education | Follow-up Knowledge-based Education
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 10 | 6
units on a scale | 6.60 (1.88) | 6.80 (2.59) | 8.49 (2.05) | 6.93 (2.51) | 8.80 (1.87) | 6.00 (2.10)

ADVERSE EVENTS:
Arm/Group | Health Belief Model Based Education | Knowledge-based Education
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

LIMITATIONS AND CAVEATS:
Overall limitation of the trial were due to attrition at the one month follow up.

This was due to the end of school year.This meant that students were busy preparing for finals, starting co-ops/internships, moving back home, or lack of interest.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less